CLINICAL TRIAL: NCT07123025
Title: Outcome of Partial Pulpotomy in Moderate and Severe Pulpitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Prerna Yadav
Record Dates: First submitted 2025-06-23; First posted 2025-08-14 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Moderate Pulpitis; Severe Pulpitis; Extremely Deep Caries
Keywords: partial pulpotomy
MeSH Terms: conditions — Pulpitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Partial Pulpotomy in Moderate Pulpitis (Experimental): Partial Pulpotomy will be performed after establishing a clinical diagnosis of moderate pulpitis i.e. if the tooth showed symptoms triggered by cold stimuli or percussion that lasted for minutes, but pain could be stopped using medications.
  Interventions: Procedure: Partial Pulpotomy in Moderate Pulpitis
- Partial Pulpotomy in Severe Pulpitis (Active Comparator): Partial Pulpotomy will be performed after establishing a clinical diagnosis of Severe pulpitis i.e. if the tooth showed symptoms of severe spontaneous pain and clear pain reaction to warmth and cold stimuli, often, sharp to dull throbbing pain, patients have trouble sleeping because of the pain (gets worse when lying down) and tooth sensitive to touch and percussion
  Interventions: Procedure: Partial Pulpotomy in Severe Pulpitis

INTERVENTIONS:
Procedure: Partial Pulpotomy in Moderate Pulpitis — Procedure/Surgery: Outcome of partial pulpotomy in teeth with clinical signs indicative of Moderate Pulpitis.
  After caries removal and pulp exposure pulp tissue is amputated and pulpal wound will be irrigated with 3% NaOCl, and bleeding will be controlled by placing a cotton pellet soaked with 3% NaOCl over the pulpal wound for 2 to 3 minutes and will be repeated if required. Root canal therapy will be initiated in cases in which haemostasis is not achieved even after 10 minutes. Followed by capping with 2-3mm layer of MTA. A layer of RMGIC will be placed over the MTA. Then the tooth will be permanently restored with composite resin.
  Arms: Partial Pulpotomy in Moderate Pulpitis
Procedure: Partial Pulpotomy in Severe Pulpitis — Description: Procedure/Surgery: Outcome of partial pulpotomy in teeth with clinical signs indicative of Severe Pulpitis. After caries removal and pulp exposure pulp tissue is amputated and pulpal wound will be irrigated with 3% NaOCl, and bleeding will be controlled by placing a cotton pellet soaked with 3% NaOCl over the pulpal wound for 2 to 3 minutes and will be repeated if required. Root canal therapy will be initiated in cases in which haemostasis is not achieved even after 10 minutes. Followed by capping with 2-3mm layer of MTA. A layer of RMGIC will be placed over the MTA. Then the tooth will be permanently restored with composite resin
  Arms: Partial Pulpotomy in Severe Pulpitis

SUMMARY:
The aim of the study is to compare the outcome of Partial Pulpotomy in mature permanent teeth with moderate and severe pulpitis.

OBJECTIVE: Primary objective- to compare the difference in clinical and radiographic outcome of partial pulpotomy in mature permanent teeth with moderate and severe Pulpitis. Secondary objective- To evaluate and compare OHRQoL and postoperative pain after Partial Pulpotomy in teeth with Moderate Pulpitis and Severe Pulpitis. Subjects of age group 15 to 40 years will be included and divided into two groups

1. Permanent mature molars with Moderate Pulpitis
2. Permanent mature molars with Severe Pulpitis

DETAILED DESCRIPTION:
TITLE- Outcome of Partial Pulpotomy in Moderate and Severe Pulpitis It aims to answer does outcome of partial pulpotomy differ in mature permanent teeth with moderate and severe pulpitis? P (Population) - Mature permanent mandibular molars with clinical signs of irreversible pulpitis. I (Intervention) -Partial Pulpotomy in teeth with Moderate Pulpitis. C (Comparison) -Partial Pulpotomy in teeth with Severe Pulpitis. O (Outcome) -Assessment of clinical & radiographic success at 6 and 12 months follow up

-Assessment of OHRQoL & pain experience at baseline, post-operatively every 24 hours for 1 week Various studies showed partial pulpotomy is successful in managing cases of irreversible pulpitis. The word irreversible presents a problem as at least part of the pulp can be saved. As a result, Wolter's proposed a classification system based on severity of symptoms. However, the treatment modalities proposed under the classification system need to validated by further research. To the best of our knowledge, Careddu & Duncan remains the only study that has explored the success of partial pulpotomy in terms of Wolter's classification but had low numbers and uneven distribution of moderate and severe pulpitis cases. No other clinical trials were found that compared the outcomes of partial pulpotomy in cases of moderate and severe pulpitis, where ambiguity still exists regarding the best treatment modality. This study trial aims to compare the difference in clinical and radiographic outcome of partial pulpotomy in mature permanent teeth with moderate and severe pulpitis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 15-40 years.
2. Mature permanent mandibular molars with extremely deep caries on radiograph, giving positive response to pulp sensibility test.
3. For Moderate Pulpitis- strong, heightened and prolonged reaction to cold, which can last for minutes, possibly percussion sensitive and spontaneous dull pain that can be more or less suppressed with pain medication.

   For Severe Pulpitis- Severe spontaneous pain and clear pain reaction to warmth and cold stimuli, often, sharp to dull throbbing pain, patients have trouble sleeping because of the pain (gets worse when lying down). Tooth is very sensitive to touch and percussion.
4. Pulpal bleeding can be controlled within 10 minutes
5. Patients having normal periapical status with periapical index (PAI) score ≤ 2
6. Periodontally healthy teeth
7. Positive response to pulp sensibility test

Exclusion Criteria:

1. Non restorable teeth
2. Negative response to vitality testing
3. Presence of sinus tract or soft tissue swelling
4. Absence of deep carious lesions radiographically
5. Radiographic signs of internal or external root resorption
6. Patient had moderate to severe pain, but preferred root canal treatment
7. Presence of sound dentin over pulp and pulp not exposed intraoperatively
8. Pulp haemorrhage could not be arrested within 10 minutes.
9. Necrotic pulp evident upon exposure
10. Pregnant women
11. Absence of antagonist teeth

Ages: 15 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-04-18 (Actual); Primary Completion 2026-04-18 (Estimated); Study Completion 2027-04-18 (Estimated)

PRIMARY OUTCOMES:
success rate at one year | Baseline to 12 months
  Criteria for success:-
  Clinical:
  1. Absence of signs and symptoms of spontaneous pain or pain on stimulus and discomfort except for the first few days after treatment.
  2. No tenderness to palpation or percussion and the tooth is functional.
  3. Normal mobility and probing pocket depth.
  4. Absence of associated soft tissue swelling, sinus or fistula. Radiographic: -
  1. Absence of any periapical or interradicular radiolucency. 2. Complete radiographic healing (PAI score 1 or 2 acc. to Ostravik et al). 3. Absence of internal and external root resorption Tooth will be considered successful when all the above parameters are met.

SECONDARY OUTCOMES:
Postoperative Pain | Baseline and at 24 hours, Day 2, Day 3, Day 4, Day 5, Day 6 and Day 7 after the treatment
  Post Operative Pain To assess incidence and intensity of pain postoperatively at every 24 hours till 7 days using Visual analogue Scale of 0 to 100 millimeter line. Score 0 means no pain and Score100 means maximum pain. To assess incidence and intensity of pain postoperatively at every 24 hours till 7 days using Visual analogue Scale of 0 to 100 millimeter line. Score 0 means no pain and Score 100 means maximum pain.
OHRQoL assessment | Baseline and at 24 hours, Day 2, Day 3, Day 4, Day 5, Day 6 and Day 7 after the treatment
  OHIP-14 questionnare will be used to assess the quality of life.It consists of questionnaire in seven dimensions: functional limitation, physical pain, psychological discomfort, physical disability, psychological disability, social disability, and handicap. It will be scored using a Lickert scale: never=0; hardly ever=1; occasionally=2; fairly often=3; very often=4. Total score will be calculated ranging from 0-56, with higher score denoting the worst OHRQoL

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Pankaj Sangwan, MDS, Principal Investigator — PGIDS, Rohtak, Haryana 124001
Locations (1):
- PGIDS Rohtak, Rohtak, Haryana, India